CLINICAL TRIAL: NCT00004736
Title: Viral and Immune Dynamics in HIV-Infected Patients With Tuberculosis
Brief Title: Effectiveness of Anti-HIV Therapy (HAART) in HIV-Infected Patients With Tuberculosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG A5062; AACTG A5062
Record Dates: First submitted 2000-02-25; First posted 2001-08-31 (Estimated); Last update posted 2008-09-11 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Tuberculosis; Rifabutin; AIDS-Related Opportunistic Infections; Drug Therapy, Combination; Antitubercular Agents; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Tuberculosis; AIDS-Related Opportunistic Infections | interventions — Nelfinavir; Ethambutol; Isoniazid; Pyrazinamide; Lamivudine; Rifabutin; Stavudine; Zidovudine

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Ethambutol hydrochloride
Drug: Isoniazid
Drug: Pyrazinamide
Drug: Lamivudine
Drug: Rifabutin
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to see if a type of anti-HIV therapy called HAART is effective in lowering levels of HIV and boosting the immune system in HIV-infected patients with tuberculosis (TB).

HIV-infected patients with TB have higher levels of HIV and lower CD4 cell counts (cells in the body that fight infection) than HIV-infected patients without TB. HAART has been effective in reducing HIV levels and increasing CD4 cells in patients without TB. However, its effects in HIV-infected patients with TB are unknown.

DETAILED DESCRIPTION:
Previous studies have focused on characterizing viral and immune dynamics after initiation of HAART in patients without opportunistic infection. The development of TB in HIV-infected individuals is associated with an elevation in HIV RNA levels, a decrease in CD4 cell counts, and an increase in activated (CD38) lymphocytes and proinflammatory cytokines (IL-1, TNF-alpha, and IL-6). Response to HAART may differ in individuals with an active opportunistic infection such as TB.

HIV-infected patients with active TB follow an anti-TB regimen including rifabutin and are observed for a maximum of 24 weeks before they initiate HAART. Plasma samples for 24-hour post-rifabutin dosing are collected at entry and at Weeks 4, 8, and 12, then again at Weeks 2, 3, 4, 12, and 24 after HAART initiation. Analyses of these samples are used to explore the relationship between cytokines and rifabutin metabolism and the effect of nelfinavir on rifabutin pharmacokinetics. The HAART regimen is nelfinavir plus lamivudine (3TC) plus either zidovudine (ZDV) or stavudine (d4T). After initiation of HAART, all patients undergo intensive monitoring of viral and immune dynamics for 2 months. The patients continue to be followed for 1 year from the time of starting HAART. Neither the HAART drug regimen nor anti-TB medications will be provided by the study and must be obtained by prescription. If patients are intolerant of the HAART regimen or exhibit virologic rebound, primary providers can alter or modify this regimen. As part of substudy A5065s, patients who experience signs or symptoms of paradoxical reactions (i.e., new persistent fevers that develop after initiating HAART and which last for more than 1 week without an identifiable source; marked worsening or emergence of intrathoracic lymphadenopathy, pulmonary infiltrates; worsening or emergence of cervical adenopathy on serial physical examinations; or worsening of other tuberculous lesions) have additional clinical evaluations (including a chest x-ray, a target clinical assessment, concomitant medications, and signs and symptoms) weekly for 4 weeks, then every month thereafter until the symptoms resolve.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have an HIV RNA level of 20,000 copies/ml or more within 30 days of study entry.
* Are at least 18 years old.
* Agree to use an effective method of birth control during the study.
* Agree to be treated with rifabutin at least 2 weeks before starting HAART (applies only to patients infected with TB).
* Plan to start HAART within 6 months of starting TB therapy (applies only to patients infected with TB).
* Can take 3TC, nelfinavir, and either ZDV or d4T.
* Are available for follow-up for at least 1 year.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have taken a combination of anti-HIV drugs for greater than 3 months.
* Have started HAART since they were infected with TB (applies only to patients infected with TB).
* Are resistant to more than one medication used to treat TB (applies only to patients infected with TB).
* Have had more than 16 weeks of TB therapy (applies only to patients infected with TB).
* Are taking rifampin to treat TB and cannot switch to rifabutin at least 2 weeks before starting HAART (applies only to patients infected with TB).
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44

CONTACTS AND LOCATIONS:
Overall Officials: Diane Havlir, Study Chair; Constance Benson, Study Chair
Locations (10):
- United States (10):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Cook County Hosp, Chicago, Illinois
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Brown Univ / Miriam Hosp, Providence, Rhode Island
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee